CLINICAL TRIAL: NCT00296543
Title: Pilot Study of a Noninvasive Predictor of Sudden Cardiac Death in Hemodialysis Patients
Brief Title: T Wave Alternans in Hemodialysis
Status: Completed | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Allon Friedman, MD, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: 0508-02
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: End Stage Renal Disease; Coronary Heart Disease; Congestive Heart Failure
Keywords: hemodialysis; sudden cardiac death
MeSH Terms: conditions — Kidney Failure, Chronic; Coronary Disease; Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine if the hemodialysis procedure changes the risk for cardiac arrest in patients.

DETAILED DESCRIPTION:
One-third to one-quarter of hemodialysis patients die of sudden cardiac death (SCD). The hemodialysis procedure may theoretically increase the risk of SCD. This study uses T wave alternans, a noninvasive marker of SCD, to objectively determine whether the hemodialysis procedure alters the risk of SCD in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Normal sinus rhythm

Exclusion Criteria:

* Inability to give written informed consent
* Active cardiac ischemia
* Pacemaker
* Inability to perform a brief walking treadmill test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients with heart disease and/or poor cardiac function
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2005-10; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allon Friedman, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States